CLINICAL TRIAL: NCT03344991
Title: Cardboard Cot in Neonatal Thermoregulation: Prevention of Moderate or Severe Hypothermia in Preterm Infants Assigned to Open Crib
Brief Title: Cardboard Cot: Prevention of Moderate or Severe Hypothermia in Preterm Infants Assigned to Open Crib
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 019
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Infant, Premature
Keywords: Hypothermia; Newborn
MeSH Terms: conditions — Premature Birth; Hypothermia

STUDY DESIGN:
Intervention Model Description: Infants will be randomized to either open crib (standard of care) or mylar-lined cardboard box following care in a radiant warmer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardboard Cot Care (Active Comparator): Stable infant will be transferred to cardboard cot, lined with reflective film for duration of hospital stay following weaning from radiant warmer. Infant's axillary temperature will be taken at 1 hour, 6 hours, 24 hours after being placed in the cot or crib, and then once every 24 hours until discharge.
  Interventions: Other: Cardboard Cot Care
- Open Crib (Placebo Comparator): Stable infant will be transferred to standard of care open crib for duration of hospital stay following weaning from radiant warmer. Infant's axillary temperature will be taken at 1 hour, 6 hours, 24 hours after being placed in the cot or crib, and then once every 24 hours until discharge.
  Interventions: Other: Open Crib

INTERVENTIONS:
Other: Cardboard Cot Care — When ready to be weaned from radiant warmer, infant will be placed in a reflective film-lined cot for the duration of hospitalization. Axillary temperatures will be taken at 1 hour, 6 hours, and 24 hours after placement in cot, and every 24 hours thereafter until discharge. If temperatures found < 36.0 at any time, an additional blanket and hat will be added to infant to improve temperature. All other care will be standard of care at University Teaching Hospital, including early and exclusive breastfeeding, appropriate bundling, and Kangaroo Mother Care as continuously as possible.
  Arms: Cardboard Cot Care
Other: Open Crib — When ready to be weaned from radiant warmer, infant will be placed in a standard of care open crib for the duration of hospitalization. Axillary temperatures will be taken at 1 hour, 6 hours, and 24 hours after placement in cot, and every 24 hours thereafter until discharge. If temperatures found < 36.0 at any time, an additional blanket and hat will be added to infant to improve temperature. All other care will be standard of care at University Teaching Hospital, including early and exclusive breastfeeding, appropriate bundling, and Kangaroo Mother Care as continuously as possible.
  Arms: Open Crib

SUMMARY:
Infants with an estimated gestational age < 36 6/7 weeks at delivery who have been in an incubator in the newborn ICU for at least 24 hours in settings where an incubator is available, or who are delivered in a setting where an incubator is not available, will be randomized to either standard protocol of open crib or mylar-lined cardboard cot for the duration of the hospital stay. Axillary temperatures will be taken 1 hr, 6 hrs, and 24 hours after being placed in the cot or crib, and then once every 24 hours. All other care is provided as standard of care.

DETAILED DESCRIPTION:
Following parental consent, preterm infants with an estimated gestational age < 36 6/7 weeks at delivery who have been in an incubator in the newborn ICU for at least 24 hours in settings where an incubator is available, or who are in the newborn ICU in a setting where an incubator is not available, will be randomized to to transfer either standard protocol of open crib or mylar-lined cardboard cot when their temperatures are stable for transfer. The infants will remain in the cot or crib for the duration of the hospital stay. Axillary temperatures will be taken 1 hr, 6 hrs, and 24 hours after being placed in the cot or crib, and then once every 24 hours. All other care is provided as standard of care, including WHO warm chain thermoregulation guidelines of early and exclusive breastfeeding, appropriate bundling and Kangaroo Mother Care as continuously as possible.

If at any point a babies becomes moderately (32.0-35.9° C) or severely hypothermic (< 32.0° C), an extra blanket will be added to their bodies and a hat placed on their heads.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age < 36 6/7 weeks
* Hospitalized in the newborn ICU at University Teaching Hospital
* Nursed in an incubator for at least 24 hours
* Thought to be ready to be weaned from incubator by the clinical staff

Exclusion Criteria:

* Major congenital anomalies
* Requiring ongoing respiratory support
* Suspected sepsis

Ages: 24 Hours to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Moderate (32.0-35.9° C) or Severe (<32.0° C) Hypothermia at discharge per axillary Temperature | Up to 14 days

SECONDARY OUTCOMES:
Hypothermia (< 36.0° C) throughout the duration of the intervention measured by axillary temperature | Up to14 days
Mean Axillary Temperatures on All Infants Weaned to Cardboard Cots | 4 months
Mean Axillary Temperatures on All Infants Weaned to Open Cribs | 4 months
Moderate Hypothermia (32.0-35.9° C) after placement in warming device measured by axillary Temperature | 1 hour after placement in warming device
Moderate Hypothermia (32.0-35.9° C) after placement in warming device measured by axillary temperature | 6 hours
Moderate Hypothermia (32.0-35.9° C) after placement in warming device measured by axillary temperature | 24 hours after placement in warming device
Severe (<32.0° C) Hypothermia after placement in the warming device measured by axillary temperature | 1 hour after placement in warming device
Severe (<32.0° C) Hypothermia after placement in the warming device measured by axillary temperature | 6 hours after placement in warming device
Severe (<32.0° C) Hypothermia after placement in the warming device measured by axillary temperature | 24 hours after placement in warming device
Rate of Hyperthemia (>38° C) measured by axillary temperature | 14 days
Rate of Normothermia (>36.5° C) at discharge measured by axillary temperature | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, MB BCh BAO, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No